CLINICAL TRIAL: NCT01616836
Title: Optimizing Pain and Rehabilitation After Knee Arthroplasty - Randomized, Blinded Clinical Trial Comparing Continuous Femoral Nerve Block Versus Single Injection Femoral Nerve Block Versus Local Infiltration Analgesia
Brief Title: Optimizing Pain and Rehabilitation After Knee Arthroplasty
Acronym: OPRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Anesthesiologists' Society (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Dr. Stephen Choi, Staff Anesthesiologist, Associate Professor Department of Anesthesia, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 011-2012
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- continuous FNB (Active Comparator): Bolus femoral nerve block (ropivacaine 0.5% 20 mL), continuous infusion 48 hours (ropivacaine 0.2%, 5 mL/h), placebo local infiltration
  Interventions: Other: continuous FNB
- single FNB (Active Comparator): femoral nerve block (ropivacaine 0.5% 20 mL), placebo femoral nerve block infusion, placebo local infiltration
  Interventions: Other: single femoral nerve block
- LIA (Active Comparator): placebo fascia iliac block, placebo fascia iliaca infusion, local infiltration analgesia
  Interventions: Other: local infiltration analgesia

INTERVENTIONS:
Other: continuous FNB — femoral nerve block (ropivacaine 0.5%, 20 mL) with femoral nerve block infusion 48 h (ropivacaine 0.2%, 5mL/h), placebo local infiltration
  Arms: continuous FNB
Other: single femoral nerve block — single femoral nerve block (ropivacaine 0.5%, 20 mL), placebo femoral nerve block infusion, placebo local infiltration
  Arms: single FNB
Other: local infiltration analgesia — placebo fascia iliac block, placebo fascia iliaca infusion, local infiltration analgesia (tricompartmental injection of 150 mL ropivacaine 0.2%, ketorolac 30 mg, epinephrine 10 microg/mL)
  Arms: LIA

SUMMARY:
The aim of this study is to determine the best method of pain control that will help with rehabilitation after total knee arthroplasty (TKA). Currently, the best method for pain control after TKA appears to be continuous femoral nerve block (FNB) where a small tube is placed beside the nerve that provides sensation to a large part of the knee and local anesthetic infused after surgery causing numbness to the surgical site. A single injection method also exists and may provide similar benefits. Both methods require training and can result in side effects such as temporary weakness (while the local anesthetic is still working) that can inhibit rehabilitation. A newer method injecting local anesthetic into the joint after surgery (Local Infiltration Analgesia (LIA)) is becoming common, does not cause weakness and can be done quickly at the end of surgery. It is unknown if the pain control provided by LIA is as good as that of FNB. This study will compare the femoral nerve block, continuous femoral nerve block and LIA technique to determine which provides better pain relief after TKA.

DETAILED DESCRIPTION:
This will be a prospective, randomized, double blind study. Patients will be randomized using a computer-generated sequence to one of three groups:

Group 1: Continuous femoral nerve block group (cFNB) Group 2: Single injection femoral nerve block group (sFNB) Group 3: Local infiltration analgesia group (LIA)

Inclusion criteria: Patients between the ages of 18 and 85 having primary tri-compartmental total knee arthroplasty.

Exclusion criteria: Allergy, intolerance, or contraindication to any study medication (see below), inability to walk independently prior to TKA, inability to comprehend French or English, use of major tranquilizers, ASA 4 or 5, BMI > 40, opioid tolerance (opioid consumption > 30mg oral morphine or equivalent per day), pregnancy

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing primary, tri-compartmental knee arthroplasty

Exclusion Criteria:

* Allergy, intolerance, or contraindication to any study medication
* Inability to walk independently prior to TKA
* Inability to comprehend French or English
* Use of major tranquilizers
* ASA 4 or 5
* BMI > 40
* Opioid tolerance (opioid consumption > 30mg oral morphine or equivalent per day)
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale for Pain | 09h00 on postoperative day 2
  Pain at this time is the primary impediment to beginning physiotherapy and achieving discharge criteria

SECONDARY OUTCOMES:
Opioid consumption | Cumulative 4 day consumption
  Opioid consumption is a surrogate outcome for pain. A reduction in opioid consumption also confers benefits of reduced side effects - nausea, dizziness, sedation, respiratory depression
Knee range of motion | Measured each postoperative day (4 day maximum) during daily physiotherapy session
  Active and passive range of motion - physical outcome measure
Six minute walk test | Measured once at the first postoperative visit with the surgeon, 6 weeks postoperative
  Validated functional outcome measure after total knee arthoplasty
Timed up and go | Measured once on postoperative day 2 during the physiotherapy session
  Functional outcome measure
WOMAC | Baseline questionnaire given preoperatively, at first postoperative visit (6 weeks), and second postoperative visit (3 months)
  Western Ontario and McMaster University Osteoarthritis Index - functional outcome measure questionnaire
LEFS | Baseline questionnaire given preoperatively, at first postoperative visit (6 weeks), and second postoperative visit (3 months)
  Lower extremity functional scale - functional outcome questionnaire
Incidence of motor block | Participants will be followed for the duration of hospital stay, an expected average of 4 days
  weakness in quadriceps from femoral nerve block can delay physiotherapy and cause falls
Complications of femoral nerve block, local infiltration analgesia | From date of randomization until the first postoperative visit at 6 weeks
  hematoma, infection, persistent neurological deficit 6 weeks postoperatively
Inability to ambulate/falls | Participants will be followed for the duration of hospital stay, an expected average of 4 days
Nausea | Participants will be followed for the duration of hospital stay, an expected average of 4 days
NRS for pain | The highest NRS will be assessed daily during the patient's physiotherapy session, as well as the highest NRS achieved at 2 weeks, 6 weeks, and 3 months postoperatively
  Assessing worst pain during physiotherapy, later dates to assess for the incidence of chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Colin J McCartney, MBChB, Principal Investigator — Sunnybrook Health Sciences Centre; Stephen Choi, MD, Study Director — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario